CLINICAL TRIAL: NCT03382938
Title: Wound Infiltration With Dexmedetomidine in Cesarean Section: Effect on Postoperative Analgesia
Brief Title: Dexmedetomidine Wound Infiltration in Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi Matsota, Assoc Prof of Anaesthesiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WIWDICS
Record Dates: First submitted 2017-12-17; First posted 2017-12-26 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain
Keywords: dexmedetomidine; ropivacaine; wound infiltration; ceasarean section
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dexmedetomidine (Active Comparator): Drug: dexmedetomidine (Dexmed) 20 mL solution of dexmedetomidine used for wound infiltration
  Interventions: Drug: Dexmedetomidine
- Ropivacaine (Active Comparator): Drug: ropivacaine 20 mL solution of ropivacaine 0.375% used for wound infiltration
  Interventions: Drug: Ropivacaine
- Dexmedetomidine - Ropivacaine (Active Comparator): Drug: dexmedetomidine (Dexmed) combined with Drug: ropivacaine 20 mL solution of dexmedetomidine 1γ/kg within ropivacaine 0.375% used for wound infiltration
  Interventions: Drug: Dexmedetomidine - Ropivacaine
- 0.9 % saline (Placebo Comparator): Drug:0.9 % saline solution (Normal saline). 20 ml with 0.9 % saline solution used for wound infiltration
  Interventions: Other: 0,9% saline

INTERVENTIONS:
Drug: Dexmedetomidine — WOUND INFILTRATION IN CESAREAN SECTION
  Other Names: Dexmed
  Arms: Dexmedetomidine
Drug: Ropivacaine — WOUND INFILTRATION IN CESAREAN SECTION
  Other Names: Ropi
  Arms: Ropivacaine
Drug: Dexmedetomidine - Ropivacaine — WOUND INFILTRATION IN CESAREAN SECTION
  Other Names: Dexmed Ropi
  Arms: Dexmedetomidine - Ropivacaine
Other: 0,9% saline — placebo WOUND INFILTRATION IN CESAREAN SECTION
  Other Names: normal saline
  Arms: 0.9 % saline

SUMMARY:
The effects of four different wound infiltration protocols in cesarean section will be investigated on parturient' pain intensity, PCA morphine consumption given, side effects and parturient' overall satisfaction.

One group will receive for wound infiltration dexmedetomidine, the second ropivacaine, the third dexmedetomidine combined with ropivacaine, while the last one will receive normal saline (placebo group).

DETAILED DESCRIPTION:
Parturients undergoing scheduled cesarean section under combined spinal-epidural anesthesia will be included in the study. Women will be randomly allocated according to the type of the solution used for wound infiltration into one of the following four groups using the closed envelop method.

Group DEX: Following the closure of the uterine incision and the rectus fascia, 20 mL solution of dexmedetomidine 1γ/kg within Normal Saline will be infiltrated subcutaneously along the skin wound edges.

Group ROPI: Following the closure of the uterine incision and the rectus fascia, 20 mL solution of ropivacaine 0.375% will be infiltrated subcutaneously along the skin wound edges.

Group DEX-ROPI: Following the closure of the uterine incision and the rectus fascia, 20 mL solution of dexmedetomidine 1γ/kg within ropivacaine 0.375% will be infiltrated subcutaneously along the skin wound edges.

Placebo Group: Following the closure of the uterine incision and the rectus fascia, 20 ml with 0.9 % saline solution will be infiltrated subcutaneously along the skin wound edges.

In Postanesthesia Care Unit, 2 mg of morphine will be administered bolus epidurally before the removal of the epidural catheter. Postoperative analgesia will be managed with the systematic administration of intravenous paracetamol 1g x 3 /day, oral celecoxib 200mg x 2 /day and PCA morphine (1 mg/ml) (setting: bolus dose 1 ml every 7 min). The total morphine consumption 24 hours after the PCA device initiation will be recorded.

Also, ranitidine 50 mg and metoclopramide 10 mg will be given intravenously twice per day, while ondansetron 4 mg will be prescribed to be administered intravenously in case of postoperative nausea or vomiting (max x 3 times/day).

Postoperative pain will be assessed in rest and mobilization using the Visual Analogue Scale (VAS, 0-10) at 1, 3, 6, 12, 18 and 24 hours after the end of surgery from an anesthesiologist who does not know the group assignment. Also, at the same time points, hemodynamic parameters of the parturients, side effects (nausea, vomiting, sedation, pruritus) and complications (fever, infection in the area of the wound infiltration, bleeding) will be recorded, while 24 hours postoperatively the overall patient' satisfaction with her postoperative analgesia management will be assessed using a 4 point scale.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy >37 weeks, ASA I-II, BMI<35

Exclusion Criteria:

* patient refusal, epilepsy, GERD, morbid obesity, drug allergy, ASA class >2, presence of atrioventricular block, severe systemic disease, multiple gestation, high risk pregnancy, contraindications to epidural technique, a history of severe systemic disease, recreational drug or alcohol use

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 100 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Pain score | up to 24 hours after the end of surgery
  Postoperative pain will be assessed in rest and mobilization using the Visual Analogue Scale (VAS, 0-10)

SECONDARY OUTCOMES:
morphine consumption | 24 hours after the PCA device initiation will be recorded
  morphine given by PCA (1 mg/ml)(setting: bolus dose 1 ml every 7 min).
overall patient satisfaction | 24 hours after the end of surgery
  overall patient satisfaction with postoperative analgesia using a 4 point scale

CONTACTS AND LOCATIONS:
Locations (1):
- Paraskevi K Matsota, Athens, Other, Greece

IPD SHARING:
Plan to Share IPD: Undecided